CLINICAL TRIAL: NCT05907005
Title: Instant Message-delivered Early Psychological Intervention in Stroke Family Caregivers: a Mixed-method Study
Brief Title: Instant Message-delivered Early Psychological Intervention in Stroke Family Caregivers
Acronym: EPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EPI2023
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Caregiver Burden; Mobile Phone Use
Keywords: Cognitive-behavioural therapy; ecological momentary intervention; early psychological intervention
MeSH Terms: conditions — Stroke; Caregiver Burden; Cell Phone Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Receive iCBT-based EMI with message content, delivery frequency and timing personalised to participants' preferences.
  Interventions: Behavioral: iCBT-based EMI
- Control Group (No Intervention): Receive general mental health information through instant message.

INTERVENTIONS:
Behavioral: iCBT-based EMI — Consists of brief iCBT for psychological support (mandatory), stroke care education (optional), and nurse-led real-time chat-based support messages, delivered according to participants' preferences.
  Arms: Intervention Group

SUMMARY:
Psychological distress including depression and anxiety is a major component of caregiver stress, and its negative impact on caregivers' health and well-being has been established in the literature. A recent meta-analysis reported the prevalence of depression and anxiety in stroke caregivers as 40.2% and 21.4% respectively.

An evidence profile report by the World Health Organization(WHO) has emphasised that psychological support is crucial in helping caregivers in the community to continue caring for individuals with long-term disabilities, such as stroke patients. Therefore, early psychological intervention (EPI) is crucial to improve the management and prognosis of an individual who are facing stressful events like caregiving.

The main aim of this study is to prevent or alleviate the significant psychological consequences in carers resulting from stroke events in family members. Internet-delivered cognitive-behavioural therapy (iCBT) is delivered as an ecological momentary intervention (EMI) to support the clients to engage in cognitive reframing and empower them with proper knowledge, skills and attitudes to make behavioural changes.

ELIGIBILITY:
Inclusion Criteria:

* Primary family caregiver of first-ever stroke patient who has <15 modified Barthel Index(mBI) scores (moderate disability);
* Caregiver of a stroke patient who has a hospital inpatient stay of ≥6 days and ≤21days;
* Aged ≥18;
* Able to read and communicate in Chinese (Cantonese or Putonghua);
* Able to use mobile phone instant messaging function; and
* PHQ-9 (depressive symptom) score ranging from 5 to 19 (note. mild: 5-9, moderate: 10-14, moderately severe: 15-19 and severe: 20-27)

Exclusion Criteria:

* Caregiver of stroke patient who is admitted to intensive care unit;
* Professional medical personnel and/or professional carer;
* Diagnosis of psychiatric disease before stroke event or currently taking psychotropic drug including antidepressants;
* PHQ-9≥20 (we shall provide information on mental health services; if needed, we shall make the appropriate referrals); and
* Currently participating in any type of psychological intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-07-24 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms (Patient Health Questionnaire-9 [PHQ-9]) | 24-week
  A 9-item scale with score ranging from 0 to 27, higher scores indicate higher severity of depressive symptom

SECONDARY OUTCOMES:
Anxiety symptoms (Generalized Anxiety Disorder-7 [GAD-7]) | 24-week
  A 7-item scale with score ranging from 0 to 21, higher scores indicate higher severity of anxiety symptoms
Stress level (Perceived Stress Scale [PSS-4]) | 24-week
  A 4-item scale with score ranging from 0 to 16, higher scores indicate higher severity of stress
Loneliness level (UCLA Loneliness Scale [ULS-8]) | 24-week
  The total score (8 items) ranges from 8 to 32 points, with higher scores suggesting a higher degree of loneliness
Acceptance and Action Questionnaire-II (AAQ-II) | 24-week
  The total score (7 items) ranges from 7 to 49 points, with higher scores suggesting a higher degree of psychological inflexibility and experiential avoidance

CONTACTS AND LOCATIONS:
Locations (5):
- Hong Kong (5):
  - Kwong Wah Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No